CLINICAL TRIAL: NCT05696665
Title: Role of Saffron and Chamomile and Their Active Compounds in the Management of Parkinson Disease in the Context of Psychometric and Biochemical Measures
Brief Title: Role of Saffron and Chamomile in the Management of Parkinson's Disease
Acronym: SAFCHEMRxPar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Collaborators: Aga Khan University Hospital, Pakistan (Other); Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Fizzah Ali, Assistant Professor, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F.2-81/2022-GENL/104/JPMC; 9447 (Other Grant/Funding Number: HEC); Dr Saara Ahmad Muddasir Khan (Other: Aga Khan University); Dr Mahboob Alam (Registry Identifier: Karachi University)
Record Dates: First submitted 2022-12-20; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease; Neurodegenerative Diseases
Keywords: saffron; Chamomile; Parkinson; Apigenin; Crocin; Neurodegenerative disorder
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases | interventions — Chamomile extract; crocin; Apigenin

STUDY DESIGN:
Intervention Model Description: GROUP A Conventional drugs only 40 GROUP B:Conventional drugs +1000 mg chamomile 30 mg saffron in a capsule form GROUP C:GROUP C Conventional drugs +500mgApigenin +30mg Crocin 40
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): conventional therapy only
  Interventions: Other: conventional therapy
- Group B (Experimental): conventional therapy +500 mg chamomile 15 mg saffron twice daily
  Interventions: Drug: Saffron and Chamomile
- Group C (Experimental): conventional therapy +500mgApigenin +30mg Crocin once daily
  Interventions: Drug: Crocin and Apigenin

INTERVENTIONS:
Other: conventional therapy — Patients will be kept on conventional therapy and no added drugs will be given
  Arms: Group A
Drug: Saffron and Chamomile — Patients will be given saffron and chamomile in capsule formulation twice daily
  Arms: Group B
Drug: Crocin and Apigenin — Active ingredients of saffron(Crocin) and Chamomile(Apigenin) will be given in capsule formultaion once daily
  Arms: Group C

SUMMARY:
In multitudinous preclinical studies, Saffron and Chamomile are found effective in treating PD. They can mitigate the neurodegenerative progression of the disease by curtailing dopaminergic and neuronal loss and by inhibiting alpha-synuclein aggregation. They also possess antioxidant and anti-inflammatory activities. The synergism of both drugs can manage Parkinson's disease and related neurological disorders although, clinical trials are needed for further elaboration. Therefore, the purpose of the study is to evaluate the effects of Saffron and Chamomile and their active compounds in treating Parkinson's disease. This combination may change psychometric measures (MDS-Unified Parkinson's Disease Rating Scale), biomarkers (including Alpha-synuclein), and oxidative stress-related to Parkinson's disease. This combination along with conventional therapy might be beneficial in managing patients with Parkinson's disease

DETAILED DESCRIPTION:
Parkinson's disease(PD) is a distinctive clinical disorder with a multifactorial range of etiology and symptoms. This neurodegenerative disease is spreading at exponent rates. It can impact individuals enormously. As a degenerative disease, its progression can span decades. The disease has profound repercussions for caregivers and is also a socio-economic burden for society SAFFRON Saffron is a spice obtained from the stigmas of the Crocus sativus L flower, grown extensively in Iran and other parts of the world, including Greece and India. According to current data, saffron cultivation and usage date back approximately 3000 years, although the oldest records of this plant date back to the Assyrian era.

Saffron is a perennial plant that grows to a height of 10 to 30 cm. Numerous leaves branch out from the bulb's center, culminating in two to three blooms. The color is determined by the amount of lycopene and carotenoid contained inside a three-branched stigma stigma.

Saffron contains 5% fat, 5% minerals, 10% moisture , 12% protein, 63% sugars and 5% crude fiber. Stigmas contain around 150 volatile chemicals, including terpenes, and alcohol, along with their esters. Three important bioactive components in Saffron are crocin, safranal, and picrocrocin, which are responsible for Saffron's taste, unique color r. Saffron's bitter flavor is created by picrocrocin, which eventually transforms into safranal. Additionally, lycopene, zeaxanthin, carotene, vitamins including thiamine and riboflavin are active components Saffron contains about 150 compounds, however the most physiologically active are two carotenoids called crocin and crocetin .Both of these compounds have been evaluated pharmacokinetically in animal and human research. According to pharmacokinetic studies Crocin is not accessible in the bloodstream as it is after oral intake but converted to crocetin in the colon. Additionally, it may cross the blood-brain barrier and enter the central nervous system through passive transcellular diffusion, making it beneficial in neurodegenerative illnesses.

CHAMOMILE Matricaria recutita chamomilla is an annual plant native to Europe and Asia with branching, tall, and smooth stems. Apigenin, apigenin-7-O-glucoside, luteolin, and luteolin-7-O-glucoside, terpene bisabolol ,caffeic acid, farnesene, chamazulene, chlorogenic acid flavonoids (apigenin, quercetin, , patuletin and luteolin), and coumarin are the chemical components found in this plant.

Pharmacological activities German chamomile is beneficial for treating stomachaches, IBS, and sleeplessness. It has anti-inflammatory, antibacterial, and relaxing properties. Additionally, it has acaricidal effects. Several animal studies have revealed that this herb has neuroprotective,anxiolytic, antimutagenic, cholesterol-lowering, wound healing, and antidiabetic effects. Chamomile was shown to have weak antibacterial and antioxidant capabilities, but substantial antiplatelet and anticarcinoma activities in in vitro experiments.

Rationale of the study :

In various preclinical studies role of saffron and chamomile is found effective in treating Parkinson disease. Their neuroprotective and antioxidant effects are also widely known. Although, efficacy of this combination in treating Parkinson disease as a clinical trial is yet to be analyzed .Therefore, this clinical trial is designed to determine the effects of saffron and chamomile as combination in compared to approved pharmacotherapy

Aim :

To study the effects of Saffron and Chamomile in the treatment of with reference to psychometric biochemical , and Insilco measures.

HYPOTHESIS Null Hypothesis There is no beneficial effects of Saffron and chamomile in the treatment of Parkinson disease Alternative Hypothesis Saffron and chamomile have efficacy in the treatment of Parkinson disease

AIM & OBJECTIVES

1. To evaluate and compare :

* clinical efficacy of saffron and chamomile in the management of Parkinson disease.
* the effects of saffron and chamomile on plasma biomarkers in the management of Parkinson disease.
* the antioxidant effects of saffron and chamomile in the management of Parkinson disease.

ELIGIBILITY:
Inclusion Criteria:

* • All diagnosed patients aged 40-years and above of either sex will be included

  * Diagnosis will be based on the UK Parkinson Disease Society Brain Bank Clinical Diagnostic Criteria reported by neurophysicians.

Exclusion Criteria:

* • Patients with atypical Parkinsonism will be excluded.

  * Patients with uncontrolled comorbidities will also be excluded.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale | 4months
  The MDS-UPDRS can be used to evaluate various aspects of Parkinson's disease, including non-motor and motor experiences of daily living and motor complications. It includes a motor evaluation and characterizes the extent and burden of disease across various populations. All items have five response options with uniform anchors of 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.Each parkinsonian sign or symptom is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment. The maximum total UPDRS score is 199, indicating the worst possible disability from PD
Levels of Alpha-synuclein and Human Neurofilament Light | 4 months
  levels of Alpha-synuclein and Human Neurofilament Light will be measured on day 0 and last day of trial using Elisa
Level of antioxidant:Superoxide Dismutase (SOD) | 4 months
  levels of Superoxide Dismutase (SOD) will be measured on day 0 and last day of trial

SECONDARY OUTCOMES:
Incidence of treatment -Emergent Adverse Events(Safety and Evaluation) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Fizzah Ali, MBBS,MPhil, Principal Investigator — Liaquat National hospital and Medical college
Locations (1):
- Jinnah Postgraduate Medical Centre (JPMC),, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All IPD and results along with publications will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publication of the primary outcomes
Access Criteria: Data and study material will be shared6months after the completion of study and after publicationsof primary outcomes

REFERENCES:
- [Result] Rajaei Z, Hosseini M, Alaei H. Effects of crocin on brain oxidative damage and aversive memory in a 6-OHDA model of Parkinson's disease. Arq Neuropsiquiatr. 2016 Sep;74(9):723-729. doi: 10.1590/0004-282X20160131. PMID 27706421
- [Result] Haeri P, Mohammadipour A, Heidari Z, Ebrahimzadeh-Bideskan A. Neuroprotective effect of crocin on substantia nigra in MPTP-induced Parkinson's disease model of mice. Anat Sci Int. 2019 Jan;94(1):119-127. doi: 10.1007/s12565-018-0457-7. Epub 2018 Aug 29. PMID 30159851
- [Result] Inoue E, Shimizu Y, Masui R, Hayakawa T, Tsubonoya T, Hori S, Sudoh K. Effects of saffron and its constituents, crocin-1, crocin-2, and crocetin on alpha-synuclein fibrils. J Nat Med. 2018 Jan;72(1):274-279. doi: 10.1007/s11418-017-1150-1. Epub 2017 Nov 17. PMID 29147836
- [Result] Inoue E, Suzuki T, Shimizu Y, Sudo K, Kawasaki H, Ishida N. Saffron ameliorated motor symptoms, short life span and retinal degeneration in Parkinson's disease fly models. Gene. 2021 Oct 5;799:145811. doi: 10.1016/j.gene.2021.145811. Epub 2021 Jul 2. PMID 34224829
- [Result] De Monte C, Carradori S, Chimenti P, Secci D, Mannina L, Alcaro F, Petzer A, N'Da CI, Gidaro MC, Costa G, Alcaro S, Petzer JP. New insights into the biological properties of Crocus sativus L.: chemical modifications, human monoamine oxidases inhibition and molecular modeling studies. Eur J Med Chem. 2014 Jul 23;82:164-71. doi: 10.1016/j.ejmech.2014.05.048. Epub 2014 May 22. PMID 24904963
- [Result] Ghasemi Tigan M, Ghahghaei A, Lagzian M. In-vitro and in-silico investigation of protective mechanisms of crocin against E46K alpha-synuclein amyloid formation. Mol Biol Rep. 2019 Aug;46(4):4279-4292. doi: 10.1007/s11033-019-04882-9. Epub 2019 May 20. PMID 31111370
- [Result] Anusha C, Sumathi T, Joseph LD. Protective role of apigenin on rotenone induced rat model of Parkinson's disease: Suppression of neuroinflammation and oxidative stress mediated apoptosis. Chem Biol Interact. 2017 May 1;269:67-79. doi: 10.1016/j.cbi.2017.03.016. Epub 2017 Apr 4. PMID 28389404
- [Result] Siddique YH, Jyoti S. Alteration in biochemical parameters in the brain of transgenic Drosophila melanogaster model of Parkinson's disease exposed to apigenin. Integr Med Res. 2017 Sep;6(3):245-253. doi: 10.1016/j.imr.2017.04.003. Epub 2017 Apr 29. PMID 28951838
- [Result] Mohammadzadeh L, Ghasemzadeh Rahbardar M, Razavi BM, Hosseinzadeh H. Crocin Protects Malathion-Induced Striatal Biochemical Deficits by Inhibiting Apoptosis and Increasing alpha-Synuclein in Rats' Striatum. J Mol Neurosci. 2022 May;72(5):983-993. doi: 10.1007/s12031-022-01990-3. Epub 2022 Mar 10. PMID 35274200
- See also: efficacy of parkinson disease — https://pubmed.ncbi.nlm.nih.gov/35274200/
- See also: Crocin Reverses Depression-Like Behavior in Parkinson — https://link.springer.com/article/10.1007/s12035-020-01941-2